CLINICAL TRIAL: NCT01910753
Title: Feasibility Study: Physical Activity Program Associated Wtih Nutrition Therapeutic Education in Head and Neck Cancer Population Treating by Chemotherapy With or Without Radiotherapy.
Brief Title: Physical Activity Program and Nutrition Therapeutic Education During Treatment of Head and Neck Cancer Population
Acronym: APANVADS
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Not enough patients
Sponsor: University Hospital, Limoges (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: I12018 APANVADS
Record Dates: First submitted 2013-07-22; First posted 2013-07-30 (Estimated); Last update posted 2016-09-07 (Estimated); Status verified 2016-09

CONDITIONS: Neck Cancer
Keywords: Head and neck cancer,; physical activity,; nutrition therapeutic education
MeSH Terms: conditions — Head and Neck Neoplasms; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- APA (Experimental): Patient with neck cancer and accepting the physical activity program .
  Interventions: Procedure: APA

INTERVENTIONS:
Procedure: APA — A 3-month program for physical activity and diet education will be followed. An exercise specialist will supervise patients twice per week, during the first six weeks. They will also follow nutrition counselling and therapeutic education by a dietician once per week. During the last six weeks, they will just follow a guide for safe and appropriate exercise regimen. The dietician will call patient weekly during this final period.

SUMMARY:
The purpose of this study is to examine the feasibility of resistance training and physical functioning associated with nutrition therapeutic education in head and neck cancer patients, during their treatment (chemotherapy with or without radiotherapy).

DETAILED DESCRIPTION:
The loss of muscle mass (i.e., sarcopenia) has been identified as a negative prognosis descriptor, disregarding the type of cancer. It is also a predictive descriptor for treatment-related toxicity. Therefore it appears crucial to save muscle mass of patients, following an adequate physical training together with a personalised diet program. The latter point is of major importance as malnutrition concerns 45% patients having head and neck cancer cancer, who stop physical activity due to extreme tiredness and decrease of quality of life. In the present project, we plan a physical activity program that would be adapted to each patient, accompanied by the rethought diet over a 3-month period. The adapted physical activity (APA) is constituted of two aerobic stages and one resistance training stage per a week. The evaluation will then proceed at three different moments, namely (i) at T0 i.e., beginning of the program, (ii) at 3 months i.e., when the program will be stopped, and (iii) at 6 months i.e., three months after the program stop. This evaluation will include the success rate, the level of satisfaction, the physiological parameters (VO2max, muscle mass and strength, BMI) and quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Age>18 years
* Written informed consent provided before any study specific procedures
* Consent to cooperate for clinical assessments
* Affiliation to a social security regime or beneficiary of equivalent social protection
* Performance status between 0 and 2
* Squamous cell carcinoma of oral cavity, oropharynx or hypopharynx
* Stage III - IV (T1-T4, N0-N3, M)(UICC 2002)
* Indication of radiotherapy and chemotherapy post-operative or first-line metastatic chemotherapy or in inoperable condition
* Ability to understand the nature, goal and study methodology

Exclusion Criteria:

* Prior neoadjuvant chemotherapy
* timed vital capacity< 70%
* Presence of another severe pathology including:
* severe or chronic cardiac, pulmonary, renal and/or hepatic insufficiencies
* Cons-indication to physical activity practice, at discretion of the investigator
* Patient under guardianship
* Psychological, social, geographical, or familial reasons prohibiting physical activity and follow-up
* Any other primary tumor during the last 5 years
* Pregnant or nursing

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2013-05; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
feasibility of the APA with a composite outcome measure | 3 months
  The evaluation criteria for the PA program will be:
  * The success rate that will be reached if 80% of physical exercises will be performed by the patient, over the 3-month period,
  * The level of satisfaction that will be evaluated with questionnaires filled by the patient.

SECONDARY OUTCOMES:
Evaluation of the personalised diet program and the therapeutic education with a composite outcome measure. | 3 months
  The evaluation criteria for the personalised diet program and the therapeutic education will be:
  * The success rate that will be reached if 80% of requirements will be addressed by the patient,
  * The level of satisfaction that will be evaluated with questionnaires filled by the patient.

CONTACTS AND LOCATIONS:
Overall Officials: FRANCOIS Vincent, MD, Principal Investigator — Limoges UH; Sabrina FALKOWSKI, MD, Principal Investigator — CHU LIMOGES - Oncologie
Locations (2):
- France (2):
  - CHU LIMOGES - Explorations Fonctionnelles Respiratoires, Limoges, Limoges
  - CHU LIMOGES - Oncologie, Limoges